CLINICAL TRIAL: NCT02422771
Title: Effect of the Fédération Internationale de Football Association (FIFA) 11+ Injury Prevention Program on Performance & Movement Control in Young Female Athletes
Brief Title: Effect of the FIFA 11+ Injury Prevention Program on Performance & Movement Control in Young Female Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Startup 1
Record Dates: First submitted 2015-02-25; First posted 2015-04-21 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2015-12

CONDITIONS: Injury of Anterior Cruciate Ligament
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Athletes in this group will continue with their usual warm-up for the duration of the indoor soccer season.
- Intervention group (Experimental): FIFA 11+ warm-up
  Interventions: Other: FIFA 11+ warm-up

INTERVENTIONS:
Other: FIFA 11+ warm-up — A sequence of 15 exercises performed before soccer practices and games. The exercises include strength, agility, balance and motor control components and take about 15-20 minutes to perform. The intervention replaces any previous warm-up the athletes may have done.
  Arms: Intervention group

SUMMARY:
In response to high injury rates in soccer, the Fédération Internationale de Football Association (FIFA) developed an injury prevention program called the "11+". It is designed to replace a standard warm-up and takes about 20 minutes to complete. The program has proven remarkably effective in decreasing the rate of injury in soccer players. However, uptake of the 11+ has been less than desired. Adoption of the program may be increased if additional benefits can be demonstrated and the program is introduced at a younger age. The goals of this study are to (1)establish that young athletes can tolerate the program, and (2)measure the effects of the 11+ program on the physical performance of 10-12 year old girls. Three teams will be randomly assigned to the intervention group and carry out the 11+ program for the duration of the indoor soccer season. Another 3 teams will continue with their usual warm-up. Pre- and post-intervention, balance, agility, core strength and movement control will be assessed in all athletes. The investigators hypothesize that the athletes will tolerate the program well and that the intervention group will improve on the performance tests significantly more than the control group.

ELIGIBILITY:
Inclusion Criteria:

* Bonivital club level soccer athlete

Exclusion Criteria:

* any condition or injury present at pre-testing that may place the athlete at risk (e.g. sprained ankle)

Ages: 9 Years to 11 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in single leg squat score at 6 months | Baseline and 6 months

SECONDARY OUTCOMES:
Change in Landing Error Scoring System (LESS) score at 6 months | Baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Joanne L Parsons, PhD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No